CLINICAL TRIAL: NCT01904695
Title: Causal Inference Research of Resistant Hypertension Treatment With Recipe of Removing Both Phlegm and Blood Stasis in a Real World Study
Brief Title: Causal Inference Research of Resistant Hypertension Treatment With Chinese Approach in a Cohort Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: China Academy of Chinese Medical Sciences (Other)
Collaborators: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Ya YUWEN, Doctor, China Academy of Chinese Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 81202846
Record Dates: First submitted 2013-07-14; First posted 2013-07-22 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Primary Hypertension; Hypertension, Resistant to Conventional Therapy
Keywords: resistant hypertension; causal inference; a chorot study; recipe of removing both phlegm and blood stasis
MeSH Terms: conditions — Essential Hypertension; Hypertension Resistant to Conventional Therapy | interventions — Antihypertensive Agents; Sodium Chloride Symporter Inhibitors; Angiotensin-Converting Enzyme Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antihypertensive drugs & Herbs (Experimental): Thiazide diuretics and ACE inhibitor and β-blocker & Herbs for 8 weeks
  Interventions: Drug: Herbs; Drug: Antihypertensive drugs
- Antihypertensive drugs (Active Comparator): Thiazide diuretics and ACE inhibitor and β-blocker for 8 weeks
  Interventions: Drug: Antihypertensive drugs

INTERVENTIONS:
Drug: Herbs — Herbs 180ml by mouth every 12 hours for 8 weeks
  Other Names: recipe of removing both phlegem and blood stasis
  Arms: Antihypertensive drugs & Herbs
Drug: Antihypertensive drugs — Thiazide diuretics and ACE inhibitor and β-blocker in different dosage determined by the physician for 8 weeks
  Other Names: Thiazide diuretics and ACE inhibitor and β-blocker

SUMMARY:
The research of clinical effectiveness assessment is to explore the causal relationship between treatment and outcome.Accordingly, based on the effectiveness of tan-yu treatment, the research takes the Resistant Hypertension (RH) as example to study the causal inference methods under real world.

DETAILED DESCRIPTION:
Background: Syndrome differentiation is one of the substantial characteristics in Traditional Chinese Medicine (TCM) but is still lack of scientific evidence.The inference methods of causal relationship between treatment and clinial effect under real-word study may help.

Objectives: This study aims to assess the efficacy of Phlegm and Stasis Syndrome differentiation method in treating resistant hypertension and explore causal inference in the real-world study.

Research design and methods: It is a multi-center,prospective,two-arm,cohort study including 200 patients with resistant hypertension (doctors' diagnosis based on the American Heart Association criteria 2008).Essential hypertension subjects,aged 18-70 years,blood pressure >140/90mmHg even used to be on 3 or more medications for a month and diagnosed as Phlegm and Stasis Syndrome will be included.Thiazide diuretics and/or two more antihypertensive agents for 8 weeks, Chinese herbs (for synchronic treating phlegm and blood stasis) and nonpharmacological recommendations were initiated in the observational group and the control group received the same interventions without Chinese herbs.

Outcome measures: The primary outcomes will be Systolic (SBP) and Diastolic (DBP) blood pressure reductions and changes in symptoms and signs.Cardiac event and death incident will be the secondary outcomes.Possible side effects and adverse reactions arising from the treatment like diarrhea will be recorded.

Discussion: This is a rigorous methodology pilot study and 200 patients are enough to calculate sample size in later formal trial.

ELIGIBILITY:
Inclusion Criteria:

* Essential hypertension subjects, aged 18-70 years, blood pressure > 140/90 mm Hg even used to be on 3 or more medications for a month and diagnosed as Phlegm and Stasis Syndrome will be included.

Exclusion Criteria:

* Patients will be excluded for the following conditions: with secondary resistant hypertension because of other disease like renal disease or pheochromocytoma; included in other clinical trial in one month; pregnant or breast-feed or preparing for pregnancy female; combined with disease like stroke, coronary atherosclerotic heart disease, diabetes, chronic renal failure or mental disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2013-08; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Systolic (SBP) and diastolic (DBP) blood pressure reductions | Before treatment, 8 weeks during treatment

SECONDARY OUTCOMES:
Cardiac event | Before treatment, 24 weeks follow-up
Death incident | Before treatment, 24 weeks follow-up
Scores for symptoms and signs | Before treatment, 8 weeks during treatment

OTHER OUTCOMES:
Possible side effects and adverse reactions | 2 weeks, 4 weeks, 6 weeks, 8 weeks during treatment and 24 weeks follow-up
  Possible side effects and adverse reactions arising from the treatment like diarrhea will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Ya YUWEN, PhD, Study Director — China Academy of Chinese Medical Sciences
Locations (1):
- Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yuwen Y, Liu YQ, Wang YP, Dai JG, Liu DS, Wang YX, Han XJ. The add-on effect of a Chinese herbal formula for patients with resistant hypertension: study protocol for a pilot cohort study. J Integr Med. 2015 Mar;13(2):122-8. doi: 10.1016/S2095-4964(15)60162-5. PMID 25797643